CLINICAL TRIAL: NCT04518657
Title: Internet-Delivered Lifestyle Physical Activity Intervention for Cognitive Processing Speed in Multiple Sclerosis
Acronym: BIPAMS-Cog
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Robert W Motl, Professor, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022-0084; 1R01HD103812 (NIH)
Record Dates: First submitted 2020-08-10; First posted 2020-08-19 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Multiple Sclerosis
Keywords: Physical Activity; Cognition
MeSH Terms: conditions — Multiple Sclerosis; Motor Activity | interventions — Behavior Therapy; Exercise; Health

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Behavioral Intervention for Physical Activity in MS (BIPAMS) (Experimental): The current behavioral intervention consists of two primary components; an internet website and oneonone video chats with a behavioral coach.The internet website involves content delivered through interactive video courses.The interactive video courses are based on elements of social cognitive theory.Each course consists of an introduction,the primary content,and a take home message.The interactive courses include embedded,supplementary options such as videos on content and worksheets related to the topic.A pedometer is provided for tracking steps,and these steps will be entered into the website so progress can be monitored.The chats support adherence to the intervention,discussion of website material,supportive accountability,and reporting of adverse events/injuries.The chats are conducted facetoface through an online videoconferencing platform.The chats occur 7 times during the first 2 months,4 times during the second 2 months,and twice during the final 2 months of the intervention.
  Interventions: Behavioral: Behavioral Intervention for Physical Activity in MS (BIPAMS)
- Wellness for MS (WellMS) (Sham Comparator): Provides an internet website and oneonone video chats that discuss materials about self-managing multiple sclerosis (MS) consequences and health indicators through methods other than physical activity.The materials are transformations of brochures provided by the National MS Society,including Gait or Walking Problems:The Basic Facts;MS and Your Emotions;Pain:The Basic Facts; Solving Cognitive Problems;Taming Stress in MS;Food for Thought:MS and Nutrition;and Vitamins,Minerals,and Herbs:An Introduction.The delivery of the internet materials and chat sessions will occur on the same time schedule and frequency as the intervention condition,and will have a comparable time commitment. The control condition will not involve tracking steps and a pedometer with not be provided.
  Interventions: Behavioral: Wellness for MS (WellMS)

INTERVENTIONS:
Behavioral: Behavioral Intervention for Physical Activity in MS (BIPAMS) — A behavioral intervention that involves an internet website and one-on-one video coaching calls for increasing physical activity in people with MS.
  Arms: Behavioral Intervention for Physical Activity in MS (BIPAMS)
Behavioral: Wellness for MS (WellMS) — A behavioral intervention that involves an internet website and one-on-one video coaching calls for increasing wellness in people with MS.
  Arms: Wellness for MS (WellMS)

SUMMARY:
We propose a highly-informed, well-designed randomized controlled trial (RCT) that is critical for providing Class I evidence regarding an Internet-delivered physical activity (PA) intervention as a behavioral approach for managing slowed cognitive processing speed (CPS; the most common and perhaps most burdensome MS-related cognitive impairment) and its second learning and memory, symptomatic, and quality of life (QOL) correlates among fully-ambulatory persons with multiple sclerosis (MS) who present with CPS impairment. Such an approach will involve a single-blind, RCT that examines the effects of a remotely-delivered, Internet-based PA intervention compared with an active control condition for yielding immediate and sustained improvements in CPS, learning and memory, symptomatic, and QOL outcomes among persons with mild MS-related ambulatory impairment who demonstrate impaired CPS. The primary outcome is the raw (unadjusted), oral Symbol Digit Modalities Test (SDMT) score as a neuropsychological measure of CPS, and this will be collected remotely via screen-sharing technology. The secondary outcomes include an objective neuropsychological measure of learning and memory (California Verbal Learning Test-II) collected remotely via screen-sharing technology, self-report measures of fatigue (Fatigue Severity Scale), depressive symptoms and anxiety (Hospital Anxiety and Depression Scale), pain (Short-Form, McGill Pain Questionnaire) and QOL (Multiple Sclerosis Impact Scale-29) that will be captured remotely using Qualtrics. The tertiary outcome is accelerometry as an objective, device-based measure of steps/day that will be delivered and returned via pre-paid, pre-addressed envelopes through the United States Postal Service for generating a minimal clinically important difference value that guides the prescription of free-living PA for managing CPS impairment in clinical practice.

DETAILED DESCRIPTION:
Cognitive impairment is prevalent, disabling, and poorly-managed among the 1 million Americans living with multiple sclerosis (MS). Indeed, 67% of adults with MS have cognitive impairment, particularly slowed cognitive processing speed (CPS), and this is associated with impaired learning and memory and worse fatigue, depression, anxiety, pain, and quality of life (QOL). This underscores the importance of identifying efficacious approaches for managing CPS impairment and its consequences among those with MS. There is merit in a remotely-delivered physical activity (PA) intervention for managing MS-related CPS dysfunction in MS. We have provided evidence from a pilot, randomized controlled trial (RCT) that an Internet-delivered PA intervention resulted in a clinically meaningful improvement in CPS among those with mild MS-related ambulatory disability; there were additional improvements in fatigue, depression, anxiety, pain, and QOL. The pilot RCT did not a priori recruit persons with MS who had objective CPS impairment nor examine sustainability of CPS changes over time, and it involved a waitlist control that did not account for the effects of attention and social contact. We leverage our experiences and preliminary results, and propose an appropriately-powered, Phase-II, RCT of a highly-developed and refined Internet-delivered PA intervention focusing on walking during ambulatory activities of daily living (steps/day) for yielding immediate and sustained improvements in remotely-assessed CPS among persons with mild MS-related ambulatory disability who demonstrate impaired CPS. The proposed study, if successful, will provide Class I evidence regarding the efficacy of a 6-month, Internet-delivered, PA intervention compared with an active control condition for improving important outcomes in 300 adults with MS who present with both mild MS ambulatory disability and impaired CPS. The primary outcome is the remotely-delivered Symbol Digit Modalities Test as a measure of CPS; the secondary outcomes include a remotely-delivered, objective measure of learning and memory and self-reports of fatigue, depression, anxiety, pain, and QOL; the tertiary outcome is accelerometry as an objective, device-based measure of PA. The conditions will be delivered by persons who are uninvolved in screening, recruitment, random assignment, and outcome assessment. We will collect outcomes on 3 occasions over a 12-month period (i.e., pre-intervention, immediately post-intervention, and 6-month follow-up). The outcomes will be collected using a blinded assessor. Data analyses will involve intent-to-treat principles, and mixed-effects models and logistic regression. The proposed research may yield "real-world" guidelines for free-living PA change that can be implemented for the treatment of CPS impairment in MS. Such an opportunity for rehabilitation of cognitive function using an approach with broad reach and scalability is paramount considering the prevalent, disabling, and poorly-managed nature of CPS impairment in MS and limited resources for its treatment.

ELIGIBILITY:
Inclusion Criteria:

* Residing in the United States (residing in Alabama is not required)
* English as primary language
* Between 18+ years old
* Diagnosis of MS
* Relapse free in the past 30 days
* Internet and email access
* Currently physically inactive (GLTEQ)
* Able to ambulate without assistance (self-report and PDDS)
* Willingness to complete the questionnaires
* Willingness to wear the accelerometer
* Willingness to undergo random assignment (BIPAMS or WellMS)

Exclusion Criteria:

* Individuals not meeting above inclusion criteria
* Individuals with moderate to high risk for contraindications of possible injury or death when undertaking strenuous or maximal exercise (PARQ)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Cognition | Changes in cognition scores from Baseline, 6-Month, and 12-Month
  Symbol Digit Modalities Test (SDMT); scoring involves summing the correct number of substitutions within the 90 second interval (max = 110), higher score indicates better outcomes.

SECONDARY OUTCOMES:
Fatigue Severity | Changes in fatigue from Baseline, 6-Months, and 12-Months
  Fatigue Severity Scale (FSS); scores range between 1 (min) and 7 (max), higher scores reflect greater fatigue severity.
Fatigue Impact | Changes in fatigue from Baseline, 6-Months, and 12-Months
  Modified Fatigue Impact Scale (MFIS); scores range between 0 (min) and 84 (max), higher scores indicate greater impact of fatigue on a patient's activities.
Depressive Symptoms | Changes in depressive symptoms from Baseline, 6-Month, and 12-Month
  Hospital Anxiety and Depression Scale (HADS); scores range between 0 (min) and 21 (max), higher scores reflect greater frequency of anxiety and depressive symptoms.
Anxiety | Changes in anxiety symptoms from Baseline, 6-Month, and 12-Month
  Hospital Anxiety and Depression Scale (HADS); scores range between 0 (min) and 21 (max), higher scores reflect greater frequency of anxiety and depressive symptoms.
Quality of Life (QOL) | Changes in quality of life from Baseline, 6-Month, and 12-Month
  Multiple Sclerosis Impact Scale (MSIS-29); scores range between 0 (min) and 100 (max), higher scores indicate greater impact of disease on daily function (i.e. worse outcomes).

OTHER OUTCOMES:
Accelerometry | Changes in accelerometry data from Baseline, 6-Month, and 12-Month
  Device-based measure of physical activity and sedentary behavior (ActiGraph)

CONTACTS AND LOCATIONS:
Overall Officials: Robert W Motl, PhD, Principal Investigator — University of Illinois at Chicago
Locations (1):
- University of Illinois at Chicago, Chicago, Illinois, United States

REFERENCES:
- [Derived] Motl RW, Sandroff BM, Benedict RHB, Aldunate R, Cutter G, Barron E. Internet-delivered lifestyle physical activity intervention for cognitive processing speed in multiple sclerosis. Contemp Clin Trials. 2024 Mar;138:107446. doi: 10.1016/j.cct.2024.107446. Epub 2024 Jan 17. PMID 38242351